CLINICAL TRIAL: NCT03163667
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study Comparing CB-839 in Combination With Everolimus (CBE) vs. Placebo With Everolimus (PboE) in Patients With Advanced or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: CB-839 With Everolimus vs. Placebo With Everolimus in Participants With Renal Cell Carcinoma (RCC)
Acronym: ENTRATA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX-839-005
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: advanced, metastatic RCC; RCC; CB-839; Everolimus; CBE; Glutaminase Inhibitor; Glutaminase; Tumor Metabolism; Glutamine
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — CB-839; Everolimus

STUDY DESIGN:
Intervention Model Description: This is a double blinded placebo-controlled study where participants will be randomized 2:1 to either CB-839 plus everolimus (CBE) or placebo plus everolimus (PboE)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CB-839 + Everolimus (Active Comparator): CB-839 is administered as oral tablets twice daily (BID) in combination with standard daily (QD) everolimus in 28 day cycles.
  Interventions: Drug: CB-839; Drug: everolimus
- Placebo + Everolimus (Placebo Comparator): Placebo is administered as oral tablets BID in combination with standard QD everolimus in 28 day cycles.
  Interventions: Drug: Placebo; Drug: everolimus

INTERVENTIONS:
Drug: Placebo — oral tablets
  Arms: Placebo + Everolimus
Drug: CB-839 — oral tablets
  Other Names: telaglenastat
  Arms: CB-839 + Everolimus
Drug: everolimus — oral tablets
  Other Names: Afinitor

SUMMARY:
The primary objective of this study is to compare the progression-free survival (PFS) of participants treated with telaglenastat and everolimus versus placebo and everolimus for advanced or metastatic clear cell renal cell carcinoma (ccRCC) previously treated with the following:

* At least 2 lines of therapy, including at least 1 vascular endothelial growth factor tyrosine kinase inhibitor (VEGF TKI)
* Radiographic progression of metastatic RCC must have occurred (per investigator assessment) on or after the most recent systemic therapy and within 6 months prior to cycle 1 day 1

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Score (KPS) ≥ 70%
* Estimated Life Expectancy of at least 3 months
* Documented histological or cytological diagnosis of renal cell carcinoma with a clear-cell component.
* Measurable Disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the Investigator
* Must have received at least two prior lines of systemic therapy, including at least one VEGF TKI (e.g., sunitinib, sorafenib, pazopanib, cabozantinib)

  a) Radiographic progression of mRCC must have occurred (per investigator assessment) on or after the most recent systemic therapy and within 6 months prior to Cycle 1 Day 1 (C1D1).
* Prior treatment with other anti-cancer therapies including cytokines, monoclonal antibodies, immunotherapies, and cytotoxic chemotherapy is allowed

Exclusion Criteria:

* Prior treatment with mammalian target of rapamycin (mTOR) inhibitors (everolimus or temsirolimus) or CB-839
* Receipt of any anticancer therapy within the following windows before randomization:

  * TKI therapy within 2 weeks or 5 half-lives, whichever is longer
  * Any type of anti-cancer antibody within 4 weeks
  * Cytotoxic chemotherapy within 4 weeks
  * Investigational therapy within 4 weeks or 5 half-lives, whichever is longer
  * Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before randomization. Patients with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Unable to receive medications orally (PO) or any condition that may prevent adequate absorption of oral study medication
* Major surgery within 28 days prior to randomization
* Patients with active and/or untreated central nervous system (CNS) cancer are not eligible. Patients with treated brain metastasis must have 1) documented radiographic stability of at least 4 weeks duration demonstrated on baseline contrast-enhanced CNS imaging (eg contrast-enhanced magnetic resonance imaging [MRI] of the brain) prior to randomization and 2) must be symptomatically stable and off steroids for at least 2 weeks before randomization.
* Requirement for continued proton pump inhibitor after randomization
* Chronic treatment with corticosteroids or other immunosuppressive agents except (i) inhaled or topical steroids or replacement dose corticosteroids equivalent to ≤ 10 mg prednisone and (ii) patients receiving physiological doses of hydrocortisone for adrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Whiting, Study Director — Calithera Biosciences
Locations (38):
- United States (38):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, Rogers, Arkansas
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - Florida Cancer Specialists- South, Fort Myers, Florida
  - Florida Cancer Specialists- North, St. Petersburg, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Ochsner Clinical Foundation, New Orleans, Louisiana
  - Anne Arundel Medical Center Oncology and Hematology, Annapolis, Maryland
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Mercy Clinic Oncology & Hematology, Joplin, Missouri
  - SCRI HCA Midwest, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - North Shore Hematology Oncology Associates PC DBA NY Cancer and Blood Specialists, East Setauket, New York
  - NYU Winthrop Hospital - Cancer Clinical Trials Oncology/Hematology, Mineola, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ann B. Barshinger Cancer Institute / Lancaster General Hospital, Lancaster, Pennsylvania
  - Monongahela Valley Hospital, Monongahela, Pennsylvania
  - Charleston Hematology Oncology Associates,PA, Charleston, South Carolina
  - UT/Erlanger Oncology & Hematology, Chattanooga, Tennessee
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179
- [Derived] Lee CH, Motzer R, Emamekhoo H, Matrana M, Percent I, Hsieh JJ, Hussain A, Vaishampayan U, Liu S, McCune S, Patel V, Shaheen M, Bendell J, Fan AC, Gartrell BA, Goodman OB, Nikolinakos PG, Kalebasty AR, Zakharia Y, Zhang Z, Parmar H, Akella L, Orford K, Tannir NM. Telaglenastat plus Everolimus in Advanced Renal Cell Carcinoma: A Randomized, Double-Blinded, Placebo-Controlled, Phase II ENTRATA Trial. Clin Cancer Res. 2022 Aug 2;28(15):3248-3255. doi: 10.1158/1078-0432.CCR-22-0061. PMID 35576438

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Everolimus: Placebo oral tablets twice daily (BID) in combination with standard once daily (QD) everolimus in 28 day cycles.
- CB-839 + Everolimus: CB-839 oral tablets BID in combination with standard QD everolimus in 28 day cycles.
Period: Overall Study
Arm/Group | Placebo + Everolimus | CB-839 + Everolimus
Started | 23 | 46
Completed | 0 | 0
Not Completed | 23 | 46
Not completed — Death | 15 | 27
Not completed — Study terminated by sponsor (after primary endpoint was met) | 8 | 19

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Everolimus: Placebo oral tablets BID in combination with standard QD everolimus in 28 day cycles.
- Total: Total of all reporting groups
Arm/Group | Placebo + Everolimus | CB-839 + Everolimus | Total
Number analyzed (Participants) | 23 | 46 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.38) | 65.8 (9.18) | 64.6 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 20 | 37 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 19 | 43 | 62
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 21 | 41 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of documented disease progression (assessed by Investigator per Response Evaluation Criteria in Solid Tumors [RECIST] v1.1) within 2 scheduled scan intervals following previous evaluable radiologic tumor assessment or death for any cause, whichever occurred first. Participants with no documentation of disease progression or death on-study were censored at the date of last available tumor assessment.
  Progressive Disease (PD) per RECIST 1.1: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: As of the primary data cutoff date of 26 Apr 2019; maximum duration of follow-up for PFS was 11.2 months.
Population: Intent to Treat Population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Everolimus | CB-839 + Everolimus
Number analyzed (Participants) | 23 | 46
months | 1.91 [1.87 to 8.28] | 3.81 [2.40 to 7.43]
Statistical Analysis 1: Comparison: Placebo + Everolimus vs CB-839 + Everolimus; Stratified analysis. Stratification factors were Memorial Sloan Kettering Cancer Center (MSKCC) Prognostic Risk (favorable versus intermediate/poor risk) and number of prior therapies with a tyrosine kinase inhibitor (TKI; 1 versus > 1). Due to stratification cells having < 10 events, TKI stratification factor was removed for analysis; Test type: Superiority; p = 0.07905, Log Rank — One-sided p-value comparing the treatment groups was based on a stratified log-rank test with alternative hypothesis of survival functions being not equal; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.34 to 1.20] — Hazard ratio comparing treatment groups (experimental over control) is based on a Cox proportional hazards model. A hazard ratio < 1 favors CB-839+Everolimus (CBE), and a hazard ratio > 1 favors Placebo+Everolimus (PboE)
Statistical Analysis 2: Comparison: Placebo + Everolimus vs CB-839 + Everolimus; Unstratified analysis; Test type: Superiority; p = 0.1184, Log Rank — One-sided p-value comparing the treatment groups was based on an unstratified log-rank test with alternative hypothesis of survival functions being not equal; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.37 to 1.28] — Hazard ratio comparing treatment groups (experimental over control) is based on a Cox proportional hazards model. A hazard ratio < 1 favors CBE, and a hazard ratio > 1 favors PboE

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death from any cause. Participants with no documentation of death on-study were censored at the date at which they were last known to be alive.
Time Frame: As of the data cutoff date of 30 Sep 2020; maximum duration of follow-up for OS was 30.4 months.
Population: ITT Population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Everolimus | CB-839 + Everolimus
Number analyzed (Participants) | 23 | 46
months | 9.72 [8.21 to 25.43] | 14.37 [7.89 to NA] — The upper bound of 95% CI is not estimable because almost 41% of participants in this arm were censored.
Statistical Analysis 1: Comparison: Placebo + Everolimus vs CB-839 + Everolimus; Stratified analysis: Stratification factors are MSKCC Prognostic Risk (favorable vs intermediate/poor risk) and number of prior therapies with a TKI (1 vs > 1). Due to stratification cells having < 10 events, TKI stratification factor was removed for analysis; Test type: Superiority; p = 0.4801, Log Rank — P-value comparing the treatment groups is based on a stratified log-rank test with alternative hypothesis of survival functions being not equal; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.42 to 1.50] — Hazard ratio based on a Cox proportional hazards model. A hazard ratio < 1 favors CBE, and a hazard ratio > 1 favors PboE
Statistical Analysis 2: Comparison: Placebo + Everolimus vs CB-839 + Everolimus; Unstratified analysis; Test type: Superiority; p = 0.5603, Log Rank — P-value comparing the treatment groups is based on an unstratified log-rank test with alternative hypothesis of survival functions being not equal; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.44 to 1.56] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through the end of treatment plus 28 days. The mean duration of exposure of CB-839 was 161.3 days and the mean duration of exposure for placebo was 176.2 days.
Arm/Group | Placebo + Everolimus | CB-839 + Everolimus
All-Cause Mortality (participants affected / at risk) | 15/23 | 27/46
Serious Adverse Events (participants affected / at risk) | 8/23 | 21/46
Other Adverse Events (participants affected / at risk) | 23/23 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Everolimus (N=23) | CB-839 + Everolimus (N=46)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 5
Paraesthesia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Gait disturbance (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Everolimus (N=23) | CB-839 + Everolimus (N=46)
Diarrhoea (Gastrointestinal disorders) | 11 | 10
Nausea (Gastrointestinal disorders) | 4 | 14
Stomatitis (Gastrointestinal disorders) | 7 | 10
Abdominal pain (Gastrointestinal disorders) | 3 | 9
Vomiting (Gastrointestinal disorders) | 4 | 8
Constipation (Gastrointestinal disorders) | 2 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 12 | 22
Oedema peripheral (General disorders) | 5 | 12
Mucosal inflammation (General disorders) | 2 | 7
Chills (General disorders) | 1 | 6
Pyrexia (General disorders) | 3 | 3
Asthenia (General disorders) | 0 | 4
Pain (General disorders) | 1 | 3
Malaise (General disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 4 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 15
Leukopenia (Blood and lymphatic system disorders) | 2 | 6
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 1 | 7
Dizziness (Nervous system disorders) | 3 | 3
Tremor (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 3
Blood creatinine increased (Investigations) | 8 | 15
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 4 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 5
Weight decreased (Investigations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Pneumonia (Infections and infestations) | 2 | 3
Rash pustular (Infections and infestations) | 4 | 1
Sinusitis (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 2 | 0
Photophobia (Eye disorders) | 3 | 10
Lacrimation increased (Eye disorders) | 3 | 0
Vision blurred (Eye disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 3 | 5
Agitation (Psychiatric disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 5
Haematuria (Renal and urinary disorders) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 5
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by the PI before either a multi-site publication or 18 months after final multi-site study report. PI can only publish their own results and provide 45 days in advance notice. PI must delete any Calithera confidential information from the publication other than study results and give good faith consideration to other comments made by Calithera. The PI must delay the publication for up to 45 days if requested by Calithera and publicly acknowledge Calithera and Pfizer support.

DOCUMENTS (2):
  • Study Protocol (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT03163667/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03163667/SAP_001.pdf